CLINICAL TRIAL: NCT06870240
Title: A Randomised, Double-blind, Placebo-controlled Phase 2a Pilot Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONP-002 in Adults With Mild Traumatic Brain Injury
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oragenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONP-002-AU-001
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Mild Traumatic Brain Injury, Concussion
Keywords: concussion, traumatic brain injury, biomarkers, cognition, visual-motor
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: ONP-002, is a novel neurosteroid shown to reduce inflammation in the brain. The drug is a non-natural synthetic enantiomer given as an intranasal powder to increase availability of the therapeutic to the brain after traumatic brain injury.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized and blinded parallel study with a placebo and treatment arm at a ratio of 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 92mg of Hydroxy-propyl beta-cyclodextrin as a spray-dried powder (Placebo Comparator): The placebo is 92mg of Hydroxy-propyl beta-cyclodextrin as a spray-dried powder
  Interventions: Drug: Neurosteroid enantiomer
- ONP-002 treatment (Active Comparator): ONP-002 is 8mg API and 92 Hydroxy-propyl beta-cyclodextrin as a spray-dried powder
  Interventions: Drug: Neurosteroid enantiomer

INTERVENTIONS:
Drug: Neurosteroid enantiomer — A non-natural synthetic neurosteroid enantiomer considered a new chemical entity

SUMMARY:
This is a Phase IIa, randomized, double-blind, placebo-controlled pilot study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ONP-002 in adults with mild traumatic brain injury (mTBI).

Broadly, a mTBI, often referred to as a concussion, is a type of head trauma that causes temporary disruption to brain function, usually resulting from a blow to the head, fall, or sudden movement, and is often characterised by symptoms of headache, dizziness, confusion, memory problems, and difficulty concentrating, without significant loss of consciousness or structural brain damage on imaging tests.

The study will enroll up to 40 participants into 2 parallel treatment arms, of 20 patients each, who will receive either 16 mg (8 mg twice daily [BID]) intranasal (IN) ONP-002 or placebo, at 8-12-hour intervals consecutively for 5 days with a total of up to 9 doses.

DETAILED DESCRIPTION:
Up to 40 participants will be randomized 1:1 to receive either ONP-002 or placebo, using a block randomization algorithm.

* Control Arm: Placebo
* Interventional Arm: 8 mg BID ONP-002 (a demethylated analogue of the enantiomer of progesterone) Intranasal Participants will receive BID doses of 8 mg ONP-002 or placebo for 5 consecutive days with a total of up to 9 doses, through IN administration.

If participants receive their first dose on the morning of Day1, they will receive a total of 9 doses. If participants receive their first dose on the evening of Day 1, they will receive a total of 8 doses. The last dose of study drug for all participants will be administered in the morning on Day 5.

Objectives Endpoints To determine the feasibility of administering ONP-002 in acute mTBI patients within 12 hours of injury. • Time to enrolment post injury and first treatment with ONP-002 To investigate the safety and tolerability of multiple IN doses of ONP-002 in patients with mTBI. • Incidence and severity of AEs

* Changes in vital sign measurements
* Changes in clinical laboratory results
* Changes in ECG parameters
* Change from baseline in macroscopic nasal examination findings To measure levels of ONP-002 in plasma following multiple IN doses in patients with mTBI. • Plasma concentrations of ONP-002
* Accumulation ratio (RAUC, and RCmax) To establish POC that IN ONP-002 administration within 12 hours of injury results in blood biomarker/functional changes consistent with the proposed mechanism of action. • Changes in blood biomarker and functional scores (clinical improvement over time) from baseline in ONP-002 treated participants compared to placebo.

To establish a reproducible protocol for the combination of IN ONP-002 dosing and blood biomarker draws in mTBI patients for up to 5-days post-injury by;

* Establishing if blood biomarkers can be used as a surrogate efficacy endpoint for mTBI that could be used in later phase studies. • Correlation between blood biomarkers and patient reported outcomes, cognitive performance, and visual motor performance
* Assess correlation of the below scores with initial positive blood biomarker findings prior to first dose:

  * Post-traumatic amnesia (PTA)
  * Brief loss or alteration of consciousness (LOC and AOC)
  * Standardised Assessment of Concussion (SAC) scores Screening
* Medical history
* Prior medication use
* Height and weight
* Demographics (including age, race, sex, and ethnicity)
* Pregnancy test
* Computed Tomography (CT) Scan
* Blood Glial fibrillary acidic protein (GFAP)
* GCS
* Neurological assessment checklist (LOC, PTA, AOC)
* Neurological assessment signs and symptoms checklist Safety and Tolerability
* Concomitant medication use
* Physical examination
* Adverse event monitoring
* Vital signs (systolic and diastolic blood pressure, pulse rate, temperature, respiration rate)
* 12-lead electrocardiogram (ECG)
* Clinical laboratory safety assessments (haematology, serum chemistry, coagulation and endocrinology)
* Macroscopic nasal examination Pharmacodynamics

Blood samples will be collected throughout the study for analysis of ONP-002 levels, and mTBI biomarkers including (but not limited to):

* GFAP
* Neurogranin
* ST2 (soluble interleukin 1 receptor-like 1) Efficacy

Efficacy endpoints will include the following assessment of patient reported symptom severity and clinical assessments of cognitive and visual-motor integrity:

* Rivermead Post-Concussion Questionnaire (RPQ)
* 5-minute DANA neurocognitive battery
* King-Devick (K-D) 3-minute visual motor test
* 10 and 30-day functional status evaluation using the Glasgow Outcome Scale - Extended (GOS-E) Safety and Tolerability The number of treatment-emergent AEs (TEAEs) as well as the number and percentage of participants with at least one TEAE, will be summarized by Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term and tabulated for each dose group. Summaries of TEAEs by severity and relationship will also be presented. Summaries will also be presented for TEAEs leading to death, serious TEAEs and for TEAEs leading to study withdrawal.

Observed values and changes from baseline in vital signs (including oxygen saturation levels), macroscopic nasal examination, pulmonary function, ECG parameters and continuous clinical laboratory parameters will be summarized at each scheduled timepoint by dose group using descriptive statistics (n, mean, standard deviation, minimum, maximum, median). Categorical clinical laboratory data will be summarized at each scheduled timepoint using participant counts and percentages and tabulated by dose group. Abnormalities in clinical laboratory parameters and ECG parameters QTcF will be tabulated by dose group showing participant counts and percentages.

Physical examination findings will be listed only. Pharmacodynamics Individual participant blood biomarker concentrations at each timepoint will be listed and summarized by treatment using descriptive statistics (n, mean, standard deviation, coefficient of variation, minimum, maximum, median, and geometric mean) for each dose group.

Efficacy Observed values and changes from baseline of efficacy measures (RPQ, DANA 5-minute neurocognition test, K-D 3-minute visual motor test, GOS-E) will be summarized at each scheduled timepoint by treatment arm using descriptive statistics (n, mean, standard deviation, minimum, maximum, median).

Participants will be screened for study eligibility in the hospital Emergency Department on Day 1. Eligible participants will be transferred and confined at the clinical site until completion of post first dose assessments on Day 1 after which they will be discharged. Participants will receive a daily telephone call (reminder to administer) from clinic staff on days when they are required to self-administer at home and to complete their study diary. Study participants will then be required to attend the clinical research facility for further study assessments on Days 2, 5 and 10, and an end of study assessment on Day 30. Home nursing study assessments may be provided for participants unable to attend the clinical research facility for scheduled visits.

If participants experience any clinically significant adverse events (AEs) they may remain at the study site for further observation at the discretion of the Principal Investigator (PI).

The expected total maximum study duration for participants will be 30 days, which includes a screening on Day 1, a 5-day treatment period, and a 25-day follow-up period.

ONP-002 is being developed for the treatment of mTBI (concussion). A Phase 1 healthy adults study exploring the safety and tolerability of single and multiple ascending IN doses of ONP-002 has been completed. The current phase IIa study aims to establish that ONP-002 is safe and feasible for acute (first dose administered within 12 hours of injury) IN administration in patients with mTBI while establishing protocols for administration and proof of concept (POC) using blood biomarker panels, cognitive and visual motor assessments to be used in later phase studies.

ELIGIBILITY:
7.2.1 Inclusion Criteria

Participants with suspected concussion presenting to the emergency department will be included in the study only if they satisfy all the following criteria:

1. Participant or legal representative is willing and capable of giving written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50 kg at screening.
4. Must be diagnosed with a mTBI by all the following measures:

   * Negative CT scan for acute traumatic lesions
   * Elevated Blood Glial fibrillary acidic protein (GFAP) (≥22 pg/mL)
   * Glasgow Coma Scale (GCS) score >12
   * Neurological Signs and Symptoms Checklist with history of loss/altered consciousness
   * Neurological PTA, LOC and AOC checklist
5. Must be able to receive 1st dose of study drug within 12 hours of injury.
6. No evidence of bleeding from the nose or visual full occlusion of the nasal cavity after a macroscopic nasal examination.
7. Female patients if of childbearing potential (defined as any female who has experienced menarche and who has not undergone surgical sterilisation and is not postmenopausal):

   * Must be known to not be pregnant based on a urine or blood test prior to first dose administration.
   * Must not be breastfeeding, lactating or planning pregnancy during the study period.
   * Must agree not to become pregnant or donate ova for at least 33 days after last dose of study drug.
   * Agree to use adequate contraception (defined as use of a condom by the male partner combined with use of a highly effective method of contraception [Section 10.2.3]) from screening until at least 33 days after the last dose of study drug, if not exclusively in a same-sex relationship or abstinent as a committed lifestyle.
8. Male participants must:

   * Agree not to donate sperm from signing the consent form until at least 93 days after the last dose of study drug.
   * If engaging in sexual intercourse with a female partner who could become pregnant, must agree to use adequate contraception (defined as use of a condom combined with use of highly effective method of contraception) from signing the consent form until at least 93 days after the last dose of study drug.
   * If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, must agree to use a condom from signing the consent form until at least 93 days after the last dose of study drug.
9. Have suitable venous access for blood sampling.
10. The patient must agree to have to give their blood without ownership to the repository for blood biomarker analysis.
11. Willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

7.2.2 Exclusion Criteria

Participants will be excluded from the study if they meet any of the following criteria:

1. History or presence of other significant disorder that at the discretion of the PI or delegate is considered "serious" classifying the participant as "not a good candidate" for the study.
2. Presence of penetrating brain injury.
3. Treatment with an investigational drug in another clinical trial within 60 days or 5 half-lives of the other investigational drug (whichever is longer) prior to the first administration of study drug in this trial.
4. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

7.3 Screen Failures Participants who consent to participate in the study but fail to meet the eligibility criteria at any point during the Screening Period and until randomisation are defined as screening failures. The reason for each screening failure will be recorded on the appropriate screening and enrolment log.

7.4 Re-Screening Participants who fail screening are not permitted to be re-screened. 7.5 Participant Withdrawal Criteria

Participants will be advised that they are free to withdraw from the study at any time for any reason or, if necessary, the PI (or delegate) may discontinue a participant from the study to protect the participant's wellbeing. A participant may voluntarily withdraw or be withdrawn from the study for reasons including, but not limited to, the following:

* The need to take medication which may interfere with study measurements;
* Intolerable/unacceptable AEs;
* Noncompliance of the participant with the protocol;
* Pregnancy, as indicated in Section 12.7;
* Withdrawal of consent; or
* If, in the PI's (or delegate's) judgement, it is in the participant's best interest.

The Sponsor will be notified as soon as possible of any participant withdrawals. The date and reasons for withdrawal will be recorded in the eCRF.

Any participant who prematurely discontinues study drug, should have all scheduled assessments performed and attend all scheduled follow-up visits. If a participant withdraws or is withdrawn from the study, an attempt should be made to perform the Early Termination Visit assessments detailed in the Schedule of Assessments (SoA) in Section 1.3.

7.6 Participant Replacement Final confirmation of eligibility will be conducted prior to administration of the first dose of study drug (Day 1).

Automatic replacement of participants is allowed if a participant withdraws or is withdrawn prior to administration of the first dose of study drug.

Participants who withdraw or are withdrawn from the study after administration of the first dose of study drug for reasons other than occurrence of a treatment-related SAE, may be replaced at the discretion of the PI (or delegate) and following consultation with the Sponsor.

Any participants enrolled as replacements will be allocated to the same study treatment (treatment arm) as the participant replaced.

-

-

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Patient symptom reporting | Days 2, 5, 10 and 30 post-injurt
  Neurological questionnaires for patient symptoms including Rivermead

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia